CLINICAL TRIAL: NCT05418985
Title: The Effect of Monthly Text Message Reminder After Training on Beliefs and Practice Behaviors Regarding Women's Breast Self Examination: Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deniz Akyıldız (Other)
Responsible Party: Sponsor-Investigator, Deniz Akyıldız, Assistant Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Text Message Reminder BSE
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2021-09

CONDITIONS: Women's Breast Self Examination Beliefs; Women's Breast Self Examination Practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Women in this group were given training on breast self-examination (BSE). In the three-month period following the training, a reminder text message was sent to mobile phones by the researcher to perform BSE. The text message was sent to women with regular and regular menstrual cycles on the seventh day after the bleeding ceased, and on the first day of the month to menopausal women with irregular menstrual cycles.
  Interventions: Behavioral: Monthly reminder message about breast self-exam.
- Control droup (No Intervention): Women in this group were given training on breast self-examination (BSE). No intervention was made afterwards.

INTERVENTIONS:
Behavioral: Monthly reminder message about breast self-exam. — Monthly reminder message about breast self-exam.
  Arms: Intervention group

SUMMARY:
A randomized control trial was made to examine the effects of of monthly text message reminder after training on beliefs and practice behaviors regarding women's breast self examination.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-69,
* Able to speak and understand Turkish,
* At least primary school graduate,
* Not in pregnancy or postpartum period,
* Not in the breastfeeding process,
* Menarche,
* No current diagnosis of breast cancer,
* No breast disease that may affect the examination finding.

Exclusion Criteria:

* Those who did not complete the training on BSE,
* Those who want to leave the research,
* Those who had pregnancy during the research and
* Those who do not fill in the data forms sent to their e-mail addresses despite being reminded by message three times.

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 83 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Women's beliefs about breast self-exam levet (mean ± SD) | 3 months after BSE education
  The primary outcome of this study was the mean beliefs about breast self-exam levet (mean ± SD) of the womens at 3 months after BSE education. Women beliefs about breast self-exam level was assessed using Champion's Health Belief Model Scale.

SECONDARY OUTCOMES:
Behaviors of women performing breast self-examination | 3 months after BSE education
  The other main outcome of the study was women performing breast self-examination measured with the BSE follow-up form.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal ALKAN, Student, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey, Turkey (Türkiye)